CLINICAL TRIAL: NCT05904262
Title: The Effect of Peripheral Protective Sensation on Peripheral Muscle Strength, Functional Capacity, Balance and Physical Activity Level in Patients With Type 2 Diabetes Mellitus
Brief Title: Peripheral Protective Sensation in Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Istanbul Kent University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Melis Usul, Reserach Assistant, Istanbul Kent University
Other Study IDs: IstanbulKentU-FTR-MU-01
Record Dates: First submitted 2023-05-24; First posted 2023-06-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot; Diabetic Neuropathies
Keywords: Diabetic Foot; Diabetic Neuropathies; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetic patients: Type 2 Diabetes Mellitus. In this prospective study based on face-to-face interview method; body fat (%), skeletal muscle mass (%) (with Omron BF511 Body Composition Monitor), waist and hip circumference, lower extremity muscle strength (for quadriceps and biceps muscles) (with muscle hand held dynamometer), It is planned to measure upper extremity muscle strength (grip strength) (with hand grip dynamometer), functional capacity (with 6 Minute Walk Test), postural stability, stability limits and sensory integration of balance (with Biodex Balance System®). In addition, individuals are expected to answer the questions of the International Physical Activity Questionnaire-Short Form (IPAQ) to evaluate their physical activity levels.
  Interventions: Other: Foot Sole Sensation Evaluation

INTERVENTIONS:
Other: Foot Sole Sensation Evaluation — Type 2 Diabetes Mellitus. In this prospective study based on face-to-face interview method; body fat (%), skeletal muscle mass (%) (with Omron BF511 Body Composition Monitor), waist and hip circumference, lower extremity muscle strength (for quadriceps and biceps muscles) (with muscle hand held dynamometer), It is planned to measure upper extremity muscle strength (grip strength) (with hand grip dynamometer), functional capacity (with 6 Minute Walk Test), postural stability, stability limits and sensory integration of balance (with Biodex Balance System®). In addition, individuals are expected to answer the questions of the International Physical Activity Questionnaire-Short Form (IPAQ) to evaluate their physical activity levels.

SUMMARY:
The aim of our study was to investigate the effect of sole sensation on peripheral muscle strength, functional capacity, balance and physical activity level in individuals with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Type II diabetes mellitus (DM) is a chronic disease characterised by insulin resistance, which is common all over the world, imposes an economic burden on the patient and his/her family because it requires continuous care and treatment, and may adversely affect the quality and duration of life of patients by leading to organ and function losses due to the complications it causes. Today, diabetes is an increasingly important health problem due to its incidence and the problems it causes. In DM, macrovascular and microvascular complications are observed with the disease. It may lead to development of foot deformities, biomechanical abnormalities and loss of protective sensation in the foot due to motor, sensory and autonomic neuropathy especially in the lower extremity. In the progressive process, loss of protective sensation may result in peripheral neuropathy. In the literature, loss of protective sensation is shown as the primary cause of peripheral neuropathy. In a study, it was found that light touch pressure, two-point discrimination and vibration senses on the soles of the feet of patients with diabetes mellitus decreased compared to healthy individuals. Diabetic foot is an important complication of diabetes which can be prevented with patient education and early treatment, although mortality, morbidity and treatment costs are quite high. This condition affects the individual's life in many aspects. When reseracher examine the literature, most of the studies on physical activity, functional capacity and quality of life in individuals with Type 2 DM with neuropathy examine the effect of neuropathy on these parameters. There is little literature examining the effect of protective sensory loss before the development of neuropathy. Researcher think that it is important to evaluate the sole sensation before the development of neuropathy in type 2 DM patients in order to determine the risk factors. Researcher also think that we will contribute to the literature by examining the relationship between the level of protective sensory loss and muscle strength, functional capacity, balance and physical activity level.

The study is planned to include 30 volunteer participants diagnosed with Type 2 Diabetes Mellitus. In this prospective study based on face-to-face interview method; body fat (%), skeletal muscle mass (%) (with Omron BF511 Body Composition Monitor), waist and hip circumference, lower extremity muscle strength (for quadriceps and biceps muscles) (with muscle hand held dynamometer), It is planned to measure upper extremity muscle strength (grip strength) (with hand grip dynamometer), functional capacity (with 6 Minute Walk Test), postural stability, stability limits and sensory integration of balance (with Biodex Balance System®). In addition, participants are expected to answer the questions of the International Physical Activity Questionnaire-Short Form (IPAQ) to evaluate their physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Type 2 Diabetes Mellitus for at least 1 year
* To be between the ages of 18-65
* HbA1c value between 6.5-11
* No cognitive/mental problems
* Being able to walk independently
* Being literate in Turkish

Exclusion Criteria:

* Lack of co-operation
* Patients with uncontrolled hypertension and uncontrolled arrhythmias
* Vertigo and various vestibular system disorders
* Those with severe neurological or severe respiratory diseases
* Patients who have undergone percutaneous transluminal coronary angiography or have a cardiac pacemaker
* Previous stroke, myocardial infarction
* Patients with major musculoskeletal problems
* Chronic renal failure
* Chronic liver disease
* Patients with hip or knee replacement surgery in the last 5 years
* Patients with an injury involving the lower extremity in the last 6 months
* Those who are pregnant
* Those with haemolytic or renal anaemia
* Those who cannot read and write Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were followed up with the diagnosis of Diabetes Mellitus at the Internal Medicine Outpatient Clinic of the Eyup Additional Service Building of Bezmialem October Foundation University
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Foot Sole Sensation Evaluation | 20 minute
  Light touch pressure sensation will be assessed with the 10-g monofilament -Semmes Weinstein test. A 128 Hz diapause will be used to test the sense of vibration. Firstly, the diaposon will be applied to the patient's wrist (it can be on the elbow or clavicle), so that the patient will know what to experience beforehand. The diapozone is placed on the bone on the dorsal side of the distal phalanx of the first toe of the foot.For two-point discrimination sensation, two-point discrimination distance measurement with an esthesiometer (Baseline® , White Plains, NY, USA) will be used

SECONDARY OUTCOMES:
Body mass index | 5 minute
  Digital, portable and non-invasive "Omron BF511 Body Composition Monitor (Omron Healthcare Co.,Ltd.; Japan)" will be used to measure Body mass index (kg/m2) of the participants.
Body Fat | 5 minute
  Digital, portable and non-invasive "Omron BF511 Body Composition Monitor (Omron Healthcare Co.,Ltd.; Japan)" will be used to measure Body fat (%) of the participants.
Skeletal muscle mass | 5 minute
  Digital, portable and non-invasive "Omron BF511 Body Composition Monitor (Omron Healthcare Co.,Ltd.; Japan)" will be used to measure skeletal mass (%) of the participants.
Resting metabolism | 5 minute
  Digital, portable and non-invasive "Omron BF511 Body Composition Monitor (Omron Healthcare Co.,Ltd.; Japan)" will be used to measure resting metabolism (kcal) of the participants.
Balance | 20 minute
  Postural stability, stability limits and sensory integration of balance will be evaluated with Biodex Balance System®. Biodex Balance System® is an equipment used to evaluate postural stability, stability limits and fall risk, and validity and reliability studies have been performed
International Physical Activity Questionnaire-Short Form (IPAQ) | 3 minute
  The questionnaire includes questions about physical activity performed for at least 10 minutes in the last 7 days. In the questionnaire, it is determined how many days in the last week and how long each day was spent in heavy physical activity (VPA), moderate physical activity (MPA) and walking (W). In the last question, the time spent daily without moving is questioned.
Muscle strength | 15 minute
  The muscle strength of M. Biceps Brachii and M. Quadriceps Femoris will be performed using an electronic hand dynamometer (Commander Muscle Tester; JTECH Medical, USA). The grip force will be performed from the dominant hand using a Jamar brand dynamometer from hydraulic measuring instruments. Data obtained will be recorded in kilograms/force (kg/N)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Unıversty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No